CLINICAL TRIAL: NCT02720120
Title: A Randomized Placebo-Controlled, Multi-Center, Phase I/II Study of the Safety of Escalating Single Intravenous Doses of Ocrelizumab (rhuMAb 2H7, RO4964913, PRO70769) in Patients With Moderate to Severe Rheumatoid Arthritis Receiving Stable Doses of Concomitant Methotrexate But With Unsatisfactory Clinical Response
Brief Title: A Study of Ocrelizumab in Participants With Moderate to Severe Rheumatoid Arthritis (RA)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The overall benefit risk profile of ocrelizumab was not favorable in RA
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA18230; 2004-002132-26 (EudraCT Number)
Record Dates: First submitted 2016-03-22; First posted 2016-03-25 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (8):
- Part 1: Ocrelizumab 1000 mg (Experimental): Participants will receive single IV infusion of ocrelizumab 1000 mg.
  Interventions: Drug: Ocrelizumab
- Part 1: Ocrelizumab 1500 mg (Experimental): Participants will receive single IV infusion of ocrelizumab 1500 mg.
  Interventions: Drug: Ocrelizumab
- Part 1: Ocrelizumab 2000 mg (Experimental): Participants will receive single IV infusion of ocrelizumab 2000 mg.
  Interventions: Drug: Ocrelizumab
- Part 1: Ocrelizumab 400 mg (Experimental): Participants will receive single IV infusion of ocrelizumab 400 milligrams (mg)
  Interventions: Drug: Ocrelizumab
- Part 1: Placebo (Placebo Comparator): Participants will receive single IV infusion of placebo matched to ocrelizumab.
  Interventions: Drug: Placebo
- Part 2: Ocrelizumab 1000 mg (Experimental): Participants will receive single IV infusion of ocrelizumab 1000 mg.
  Interventions: Drug: Ocrelizumab
- Part 2: Ocrelizumab 1500 mg (Experimental): Participants will receive single IV infusion of ocrelizumab 1500 mg.
  Interventions: Drug: Ocrelizumab
- Part 2: Ocrelizumab 400 mg (Experimental): Participants will receive single IV infusion of ocrelizumab 400 mg.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Participants will receive single IV infusion of ocrelizumab at 400, 1000, 1500, and 2000 mg.
  Other Names: RO4964913, rhuMAb 2H7, PRO70769
  Arms: Part 1: Ocrelizumab 1000 mg; Part 1: Ocrelizumab 1500 mg; Part 1: Ocrelizumab 2000 mg; Part 1: Ocrelizumab 400 mg; Part 2: Ocrelizumab 1000 mg; Part 2: Ocrelizumab 1500 mg; Part 2: Ocrelizumab 400 mg
Drug: Placebo — Participants will receive single IV infusion of placebo.
  Arms: Part 1: Placebo

SUMMARY:
This study is in two parts and will evaluate the safety, tolerability and efficacy of escalating single intravenous (IV) doses of ocrelizumab compared with placebo in combination with methotrexate in participants with moderate to severe RA. Part 1 is the dose-escalation study, at one of the following dose levels of ocrelizumab [400, 1000, 1500, and 2000 milligrams (mg)]. In Part 2, participants will be randomized to explore tolerability and efficacy of doses which have been shown to be tolerated in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe RA for at least 6 months
* Positive serum rheumatoid factor (>/= 20 international units per milliliter)
* Current treatment with RA on an outpatient basis
* Treatment failure with one disease modifying anti-rheumatic drug (DMARD) or biologic, but have not failed more than six of these agents including methotrexate
* Current treatment with methotrexate for at least 12 weeks, at a stable dose
* Use of highly effective contraception.

Exclusion Criteria:

* Rheumatic autoimmune disease or inflammatory joint disease, other than RA
* Concurrent treatment with any disease-modifying anti-rheumatic drug (DMARD) (other than methotrexate) or any anti-tumor necrosis factor (TNF) -alfa or other biologic therapy
* Treatment with any other investigational drug within 4 weeks of screening
* Previous treatment with cell-depleting therapies, IV gamma-globulin, intra-articular or parenteral corticosteroids, and receipt of live/attenuated vaccine prior to screening
* Previous treatment with rituximab or any other anti-cluster of differentiation 20 (CD20) agent
* History of severe allergic or anaphylactic reactions to humanized monoclonal antibodies
* Known active bacterial, viral or fungal infections
* History of active tuberculosis and primary or secondary immunodeficiency
* History of concomitant diseases such as cardiovascular disease, nervous system, pulmonary disease, renal, hepatic, endocrine or gastrointestinal disorders
* Pregnancy or lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2005-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) or Serious AEs (SAEs) | Baseline up to approximately 7.25 years
Percentage of Participants with Anti-Ocrelizumab Antibodies | Baseline up to approximately 7.25 years

SECONDARY OUTCOMES:
Percentage of Participants with American College of Rheumatology (ACR) 20%, 50%, and 70% (ACR20/50/70) Response at Week 24 | Week 24
Disease Activity Score at Week 24 | Week 24
Percentage of Participants achieving European League Against Rheumatism (EULAR) Response at Week 24 | Week 24
Maximum Plasma Concentration (Cmax) of Ocrelizumab | Pre-infusion (0 hours); 30 minutes post infusion on Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24 (up to Week 24), and Weeks 36, 48 (Post Week 24)
Time to Blood B-Cell Depletion | Baseline up to approximately 7.25 years
Terminal Elimination Half-Life (t1/2) of Ocrelizumab | Pre-infusion (0 hours); 30 minutes post infusion on Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24 (up to Week 24), and Weeks 36, 48 (Post Week 24)
Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity AUC(0-inf) of Ocrelizumab | Pre-infusion (0 hours); 30 minutes post infusion on Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24 (up to Week 24), and Weeks 36, 48 (Post Week 24)
Area Under the Plasma Concentration-Time Curve From Time 0 to Last Quantifiable Concentration AUC(0-last) of Ocrelizumab | Pre-infusion (0 hours); 30 minutes post infusion on Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24 (up to Week 24), and Weeks 36, 48 (Post Week 24)
Time to Maximum Observed Plasma Concentration (Tmax) of Ocrelizumab | Pre-infusion (0 hours); 30 minutes post infusion on Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24 (up to Week 24), and Weeks 36, 48 (Post Week 24)
Terminal Rate Constant of Ocrelizumab | Pre-infusion (0 hours); 30 minutes post infusion on Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24 (up to Week 24), and Weeks 36, 48 (Post Week 24)
Systemic Clearance (CL) of Ocrelizumab | Pre-infusion (0 hours); 30 minutes post infusion on Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24 (up to Week 24), and Weeks 36, 48 (Post Week 24)
Mean Residence Time (MRT) of Ocrelizumab | Pre-infusion (0 hours); 30 minutes post infusion on Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24 (up to Week 24), and Weeks 36, 48 (Post Week 24)
Steady State Volume of Distribution (Vss) of Ocrelizumab | Pre-infusion (0 hours); 30 minutes post infusion on Day 1; Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24 (up to Week 24), and Weeks 36, 48 (Post Week 24)
Duration of Blood B-Cell Depletion | Baseline up to approximately 7.25 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (37):
- Australia (4):
  - Darlinghurst, New South Wales
  - Adelaide, South Australia
  - Melbourne, Victoria
  - Perth, Western Australia
- Belgium (2):
  - Ghent
  - Leuven
- Canada (6):
  - Calgary, Alberta
  - Edmonton, Alberta
  - London, Ontario
  - Toronto, Ontario
  - Québec, Quebec
  - Sherbrooke, Quebec
- Amsterdam, Netherlands
- Auckland, New Zealand
- Russia (2):
  - Moscow
  - Saint Petersburg
- Spain (9):
  - Barcelona, Barcelona
  - Cadiz, Cadiz
  - Granada, Granada
  - Santiago de Compostela, La Coruña
  - Alcorcón, Madrid
  - Madrid, Madrid
  - Seville, Sevilla
  - San Cristóbal de La Laguna, Tenerife
  - Valencia, Valencia
- United Kingdom (12):
  - Aberdeen
  - Cambridge
  - Derby
  - Leeds
  - Liverpool
  - London
  - Maidstone
  - Newcastle upon Tyne
  - Norwich
  - Salford
  - Torquay
  - West Midlands